CLINICAL TRIAL: NCT00093938
Title: Cranberry for Prevention of Bacteriuria in Pregnancy
Brief Title: Cranberry Juice for Preventing Bacteria in Urine During Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DK068527-01 (completed)
Record Dates: First submitted 2004-10-07; First posted 2004-10-08 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Urinary Tract Infection; Bacteriuria
Keywords: Vaccinium macrocarpon; Asymptomatic Bacteriuria
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

INTERVENTIONS:
Drug: Cranberry juice

SUMMARY:
The purpose of this study is to determine the amount of cranberry juice that is most effective in preventing a condition in pregnant women that often leads to urinary tract infections (UTIs).

DETAILED DESCRIPTION:
Asymptomatic bacteriuria (ASB) infection, a condition in which a large number of bacteria are present in the urine, often precedes the development of symptomatic UTIs. UTIs are common among women and may create complications during pregnancy. By incorporating cranberry juice into their diets, pregnant women may be able to lower their risk for UTIs caused by ASB, and cranberry juice may also prevent preterm labor and birth. This study will determine the cranberry juice-containing regimen that will work best for preventing ASB in pregnant women.

For the duration of their pregnancy, participants in this study will be randomly assigned to one of three treatment arms: cranberry juice once a day, cranberry juice three times a day, or a placebo beverage three times a day. The level of bacteria in their urine will be measured at monthly study visits. Women who test positive for a UTI will receive oral antibiotic therapy. All women will be monitored throughout their pregnancies for UTIs and other related complications.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy
* Mother and fetus in good health
* Mother pregnant for 16 weeks or less

Exclusion Criteria:

* Suspected nonviable or ectopic pregnancy
* Mother plans to terminate pregnancy
* Antimicrobial therapy, for reasons other than urinary tract infections, within 2 weeks prior to study start
* Significant underlying medical complications that may interfere with the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2004-12

PRIMARY OUTCOMES:
Number of cases of asymptomatic bacteriuria

SECONDARY OUTCOMES:
Number of cases of symptomatic urinary tract infection
Compliance with recommended therapy
Number of preterm deliveries

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Wing, MD, Principal Investigator — University of California, Irvine Medical Center/Long Beach Memorial Medical Center
Locations (2):
- United States (2):
  - Women's Pavilion at Miller Children's Hospital (Long Beach Memorial Medical Center), Long Beach, California
  - University of California, Irvine Medical Center, Orange, California

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Wing DA, Rumney PJ, Leu SY, Zaldivar F. Comparison of urinary cytokines after ingestion of cranberry juice cocktail in pregnant subjects: a pilot study. Am J Perinatol. 2010 Feb;27(2):137-42. doi: 10.1055/s-0029-1224867. Epub 2009 Jun 26. PMID 19562652
- [Derived] Wing DA, Rumney PJ, Preslicka CW, Chung JH. Daily cranberry juice for the prevention of asymptomatic bacteriuria in pregnancy: a randomized, controlled pilot study. J Urol. 2008 Oct;180(4):1367-72. doi: 10.1016/j.juro.2008.06.016. Epub 2008 Aug 15. PMID 18707726